CLINICAL TRIAL: NCT04227691
Title: Treatment of Axillary Hyperhidrosis With Long-pulsed Nd:YAG Laser or IPL Using Dynamic Optical Coherence Tomography Imaging of Laser-Tissue Interaction: Protocol for a Within-person Randomised Trial Conditioning on Treatment Type
Brief Title: Treatment of Axillary Hyperhidrosis With Long-pulsed Nd:YAG Laser or IPL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Gregor Jemec, Professor, PhD, DmsC, Head of Dpt., Zealand University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SJ-689
Record Dates: First submitted 2020-01-07; First posted 2020-01-14 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Hyperhidrosis Primary Focal Axilla
Keywords: localized hyperhidrosis; Nd YAG laser treatment; OCT scan; Axillary hyperhidrosis; IPL

STUDY DESIGN:
Intervention Model Description: Twenty patients are enrolled. Each patient is randomized to receive treatment in left or right axilla with either IPL or Nd:YAG. Thus, it is a within-person randomised trial, where patients receive one treatment in one axilla and the opposite axilla serve as a control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Long-pulsed Nd YAG laser treatment (Active Comparator): Ten patients will be randomized to receive Long-pulsed Nd:YAG in either left or right axilla. (The other axilla will serve as within-person control)
  Interventions: Device: Long-pulsed Nd Yag laser treatment
- IPL treatment (Active Comparator): Ten patients will be randomized to receive IPL treatment in either left or right axilla. (The other axilla will serve as within-person control)
  Interventions: Device: IPL treatment

INTERVENTIONS:
Device: Long-pulsed Nd Yag laser treatment — One treatment of the assigned axilla with long-pulsed Nd YAG laser treatment in ten patients
  Arms: Long-pulsed Nd YAG laser treatment
Device: IPL treatment — One treatment of the assigned axilla with IPL treatment in ten patients
  Arms: IPL treatment

SUMMARY:
SUMMARY Objective To assess the efficacy of Nd:YAG laser treatment on eccrine sweat production in the axillae of persons experiencing excessive axillary hyperhidrosis.

Design Randomised, within-person controlled clinical trial.

Setting One Dermatology Department, at a University hospital in Denmark, from 2018-20.

Participants A total of 10 participants enrolled after signing informed consent from the patients attending the hyperhidrosis clinic.

Interventions Participants will receive one Nd:YAG laser-treatment of either left or right axilla. The treated area will be cooled with ice during and after laser treatment. Prior to treatment, patients can use lidocaine-prilocaine 5% cream at the treatment site on an optional basis.

Main outcome measures Primary outcome measure will be reduced excessive sweat production (%points) monitored by an iodine-starch test assessed at 1-month follow-up compared to baseline. A 30% reduction in sweat production in the Nd:YAG laser-treatment relative to control, will be considered clinically significant.

Key secondary outcome measures include (1) weighing the sweat by gravimetric testing, (2) patient assessment of sweat production on a Hyperhidrosis Disease Severity Scale (HDSS) - also assessed at 1 month from baseline. Safety around the use of Nd:YAG laser-treatment will be monitored by registering pain during treatment on a visual analogue scale, as well as monitoring of adverse events immediately as well as one week after treatment. As for the purpose of further exploratory analyses (both benefits and harms), all outcome measures will be re-collected 24 months after treatment.

Timelines and dissemination For the collection of the primary data (i.e. primary endpoint being assessed after 1 month), First Patient First Visit (FPFV) will take place in November 2018 and Last Patient Last Visit (LPLV) will be in March 2019.

The investigators plan to present data internationally at e.g. the European Academy of Dermatology and Venerology as well as nationally to the Danish Dermatology Society and to the Hyperhidrosis Patient Association. Results will be published in an internationally recognised peer reviewed (biomedical) journal.

Trial registration: Danish Research Ethics Committee (approved, protocol number: SJ-689); ClinicalTrials.gov: NCT pending (2018-11-22).

DETAILED DESCRIPTION:
INTRODUCTION Primary axillary hyperhidrosis is a condition with excessive secretion of sweat from the eccrine sweat glands of the armpits that affects between 1 and 5 % of the world's population. Numbers may be underestimated since this chronical disease debuts during adolescence and is unmentionable in many cultures and social environments. Hyperhidrosis may lead to malodour and cause large sweat patches on clothes, thus affecting dressing behaviour, social activities and job opportunities. As a direct consequence, many patients experience affected psychological and social behaviour, increased mental stress and low self-esteem.

Several treatment modalities exist that may treat axillary hyperhidrosis. Systemic treatment with anticholinergic tablets is often reserved to hyperhidrosis that affects the entire body due to a substantial risk of adverse effects. Possible adverse effects (i.e. related to the intervention) include dry mouth and other mucous membranes, digestive problems, decreased ability to empty the bladder, visual disturbances and affected nervous system. Localised axillary hyperhidrosis is often treated by injections of botulinum toxin. Although this method is effective in many patients the procedure is painful, expensive and has to be repeated since the effect only last from four to nine months. Recently, heating of the sweat glands with microwave technology has shown promising efficacy with minimal adverse effects. However, this treatment is very expensive and is only available at a few sites in Denmark. Surgery has also been performed, yet short-term and long-term efficiency is inferior to other methods. Therefore, there is a need for efficient, safe, affordable and widely available alternatives to treat axillary hyperhidrosis.

An alternative method that have been proposed, could be heating and destroying sweat glands by Neodynium Yttrium Aluminium Garnet (Nd:YAG) laser or intensed pulsed light (IPL). These types of non-invasive light devices are widely available at dermatological clinics in Europe and is well-known to treat vascular lesions and undesired hair growth. The IPL has a 640 - 800 nm wavelength and the Nd:YAG laser a 1064 nm wavelength that penetrates deeply into the skin and target the melanin of the hair shaft. By adjusting the pulse length according to the theory of extended photo-thermolysis, light energy can be delivered through the hair shaft into surrounding sweat glands. A previous pilot study has demonstrated significant and lasting reduction of axillary hyperhidrosis in six patients treated with Nd:YAG laser.Treatments were reported safe and efficient without any side effects. Likewise, two studies of a comparable but invasive Nd:YAG laser technique reported only temporary mild adverse effects and significant sweat reduction for up to 43 months after treatment. A single prospective study without a control group demonstrated increased sweat production following Nd:YAG laser treatment of excessive hair growth. Targeting hair and sweat glands is however not directly comparable due to different pulse lengths of the delivered energy.

Dynamic optic coherence tomography (d-OCT) is an imaging technique that utilizes infrared light to create two-dimensional horizontal or transverse images. Penetration depth is approximately 0.5 - 2 mm 11. The d-OCT technique allows in situ visualization of dynamic changes in blood flow and superficial skin structures in vital skin. Thus, the eccrine sweat glands and the surrounding blood supply can be followed over time without taking invasive tissue biopsies. Previous studies of histological changes after laser treatment of eccrine sweat glands have only been able to demonstrate limited structural changes and therefore, there is a need for improved imaging techniques to visualize laser-tissue-interactions.

Aim & Objectives To assess the efficacy and safety of experimental intervention (either Nd:YAG laser OR IPL treatment) of an axilla with hyperhidrosis, relative to the contralateral untreated side, and to visualise laser-tissue interactions by Dynamic Optical Coherence Tomography.

Primary efficacy objective: to assess the effect of one of the experimental interventions (either Nd:YAG laser or IPL) treatment on eccrine sweat production by comparing treated and contralateral untreated axillae in patients eligible for botulinum-toxin therapy due to axillary hyperhidrosis. Sweat production is to be assessed at baseline and at one-month follow-up primarily by the iodine-starch test and secondly by gravimetric testing and questionnaires.

METHODS Patient research partners (PRPs) The study is designed without the assistance of PRPs. Collaboration between patients and professionals in developing and disseminating research projects is relatively new and the explorative nature and easily quantifiable outcomes chosen in this study reduces the need for the use of PRP. Should the study support the use of the new treatment, larger confirmatory studies will be needed and these will naturally include softer patient-rerouted outcomes and PRP collaboration.

Trial design and allocation ratio In a prospective within-person randomised trial, patients will be randomly allocated to receive laser treatment or IPL of one axilla while the other serve as a control (i.e. Right-Left and Left-Right, respectively). Primary endpoint will be assessed after 1 month. Treatments are performed with a combined platform of non-ablative 640 - 800 nm IPL and 1064 nm long-pulsed Nd:YAG laser (Lumenis M22 system, Lumenis Ltd.) and laser energy is applied according to patient skin type.

Settings and locations where the data will be collected This project will take place from autumn 2019 to spring 2021 in an established research environment in the Dermatologic Department at Zealand University Hospital Roskilde. All patients will be included from January 2020 to June 2020 and will if possible be re-evaluated two years later.

Professor, doctor in medical science and Head of Department Gregor Jemec is principal investigator. Daily leader will be medical doctor, PhD Elisabeth Hjardem Taudorf (EHT). Medical doctor and PhD-students Mattias Hennig and Linnea Thorlacius will participate in daily study activities. The department accounts for all study facilities and technical equipment. The study has been approved by the Danish Research Ethics Committee (protocol number: SJ-689). Before enrolling the first patient, the trial was registered with clinicaltrials.gov (NCT Identifier: Pending).

Interventions The intervention under investigation is one treatment with 640 - 800 nm IPL or non-ablative long-pulsed 1064 nm Nd:YAG laser (Lumenis M22 systems, Lumenis Ltd). Laser or IPL energy will be applied according to patient skin type. Skin will be cooled during and after treatment to reduce inconvenience. On an optional basis, patients may also receive topical anesthesia by lidocaine gel prior to treatment (EMLA 5%, Astra-Zenica, København S, Danmark). All patients will receive one treatment and will be followed up after one month. If possible, patients will be contacted in order to perform a long-time follow up after 24 months. After completion of the project, patients are offered laser or IPL treatment of the axilla, which served as a control in the study.

Power and Sample size considerations A sample size calculation was performed based on the assumptions that the main outcome measurement (the iodine-starch test for sweat) is continuous in nature, fairly normally distributed, and that an additional improvement in the intervention side of 30%points (assumed standard deviation=25% with a correlation of 0.5) will be considered clinically relevant. For a paired t-test of a normal mean difference with a two-sided significance level of 0.05 (p< 0.05), a sample size of 8 pairs is required to obtain a power of at least 80% to detect a mean difference between pairs of 30% (the actual power is 82.8%). It was decided to include and (within-person) randomise 10 patients for each intervention in order to consider a potential risk of drop-outs; a sample size of 10 pairs has a power of 92% to detect the mean difference between pairs of 30%.

As an extra exploratory objective, the investigators will explore whether the use of Nd:Yag laser or IPL treatment have a different outcome after assessing the overall benefit or "both of the experimental treatments". Thus, it was decided for pragmatic reasons to include 20 patients in total; 10 of them treated with Nd:Yag laser on the experimental side, whereas the other 10 will receive IPL treatment on the experimental side.

Randomization Sequence generation, allocation concealment, and implementation This is an intra-person study, comparing outcomes within participants. All participants will receive active treatment on one axilla (Active-Right|Control-Left and Control-Right|Active-Left, respectively). The implied subgroups of which axilla to receive active long-pulsed Nd:YAG treatment or IPL will also (like right/left) be selected based on a computer generated table of random numbers using SAS Proc Plan developed by an external biostatistician/author with no clinical involvement in the trial (RC). The contralateral axilla will serve as control.

The allocation will be concealed in a password-protected computer file only accessible by the biostatistician. Individual allocations will be held in sealed, opaque, consecutively numbered digital files, and forwarded individually to the principal investigator sequentially as an active feedback mechanism after receiving a scanned copy of the informed consent form. In addition, treatment of left or right axilla with either Nd:YAG or IPL will be directly communicated from the data manager to the daily leader of the project (EHT) This procedure will ensure that participants, study staff, and outcomes assessors will remain blinded to subsequent treatment allocations throughout the trial.

Statistical methods A detailed statistical analysis plan (SAP) will be developed during data collection. In brief, the analyses will be based on mixed linear models, with a random effect for participant (1, 2, 3, …, to 20) with a fixed effect for group (active or placebo), axilla (right or left), and the experimental intervention of secondary interest (Nd:YAG or IPL). For the primary analyses the type of experimental intervention (Nd:YAG or IPL) will be included as a main effect only; secondarily if the primary test hypothesis is rejected (p <0.05; H0: μActive = μPlacebo) the investigators will add a test for interaction to compare the net benefit for Nd:YAG vs. Placebo and IPL vs. placebo.

PERSPECTIVES Given a successful outcome of an investigation of long-pulsed Nd:Yag laser or IPL treatment for axillary hyperhidrosis, the laser treatment could potentially be implemented in the everyday practice, since Nd:YAG lasers and IPL devices are already widespread in European dermatological hospital departments and clinics.

Data will be presented and published internationally. This new treatment holds the potential to provide long-lasting sweat reduction in patients suffering from axillary hyperhidrosis.

Patients may benefit from improved self-esteem, prevention of social anxiety, and better job opportunities, providing a positive personal development for patients, who presently suffer from a socially unacceptable and neglected chronic disease.

ELIGIBILITY:
Inclusion Criteria:

* Legally competent
* women and men
* At least 18 years
* Fitzpatrick skin type I-III
* Suffering from severe axillary hyperhidrosis characterised by a value of 3 or 4 on the HDDS scale.

Exclusion Criteria:

* Use of photosensitizing medication
* Active treatments for axillary hyperhidrosis within the last five months.
* Wounds, scars or skin disease in the Axillae
* Prior surgery, laser or microwave therapy in the axilla
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01-17 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in sweat production measured by Iodine-starch test | from baseline to one-month post-treatment
  Reduction of sweat area measured by the percentage reduction of dark-colored area in the axilla one month after treatment measured by the iodine-starch test

SECONDARY OUTCOMES:
Change in sweat production measured by Gravimetric testing | from baseline to one-month post-treatment
  Patients sit in a calm environment at room temperature with filter pads enclosed in the axillae. The filter pads will be weighed before application to the patient and after 5 minutes to assess the amount of sweat the patient produce. A change in sweat production from baseline to one-month post-treatment will be registered.
Change in hyperhidrosis disease severity scale (HDSS) | from baseline to one-month post-treatment
  Patient's assessment at a four-point scale where 1 is barely noticeable sweat production and 4 is intolerable sweating always interfering with daily activities.
  A Change from baseline to one-month post-treatment will be registered
OCT scan of laser-tissue interactions | from baseline to one-month post-treatment
  Descriptional changes from baseline to one-month post treatment illustrated by Optical coherence tomography scan of the axillae

CONTACTS AND LOCATIONS:
Overall Officials: Gregor BE Jemec, DmSc, Prof., Principal Investigator — Zealand University Hospital - Roskilde
Locations (1):
- Zealand University Hospital Roskilde, Roskilde, Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT04227691/Prot_SAP_000.pdf